CLINICAL TRIAL: NCT06978270
Title: Healthy Start: An Innovative, Multi-level Intervention With Family Childcare Providers and Families to Improve the Dietary Behaviors of Pre-school Children
Brief Title: Healthy Start: Family Childcare Providers and Parents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK131940-01
Record Dates: First submitted 2025-03-27; First posted 2025-05-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Child Obesity; Nutrition, Healthy
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Staff who conduct evaluation in the family childcare homes will not be told which experimental condition is being provided to that home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Start: Healthy Eating in Childcare and Home Settings (Experimental): 1) Adapted version of Healthy Start nutrition intervention (peer coach using brief MI online, tailored materials, coach-led online support groups for FCCP and children's tableware and food toys for the FCCH); 2) Brief training from coach on using and scheduling healthy eating messages within the Classtag App; 3) Posters for the FCCH; 4) Tailored health eating packets (newsletters, videos and tableware/food toys) for parents.
  Interventions: Behavioral: Healthy Eating: Provider and Parent Components
- Healthy Start: Reading Readiness in Childcare and at Home (Active Comparator): An attention-matched intervention re. reading readiness and literacy promotion based on the dialogic reading technique to be delivered with a similar dose and intensity including reading readiness-focused Tailored feedback reports, monthly support coach calls, Classtag App, and tailored packets (with FCCP and parent materials) distributed monthly and online peer support groups. The FCCP will select which of the reading readiness-related and early literacy skills topics they want to work on monthly. FCCP and parents in this group will receive a set of books.
  Interventions: Behavioral: Healthy Start: Reading Readiness Childcare Proiver and Parent Materials

INTERVENTIONS:
Behavioral: Healthy Eating: Provider and Parent Components — Healthy Eating intervention for child care providers: Peer coaching using brief MI online, tailored materials, coach-led online support groups for FCCP and children's tableware and food toys; 2) Brief training on using and scheduling messages within the Classtag App; 3) Posters for the FCCH. Also for parents, healthy eating encoragement and communication from childcare providers including via the Classtag App, newsletters, videos and tableware/food toys focused on child diet at home.
  Arms: Healthy Start: Healthy Eating in Childcare and Home Settings
Behavioral: Healthy Start: Reading Readiness Childcare Proiver and Parent Materials — Reading readiness intervention for child care providers: Peer coaching using brief MI online, tailored materials, coach-led online support groups for FCCP and children's books; 2) Brief training on using and scheduling messages within the Classtag App; 3) Posters for the FCCH. Also for parents, reading readiness encoragement and communication from childcare providers including via the Classtag App, newsletters, books focused for use at home.
  Arms: Healthy Start: Reading Readiness in Childcare and at Home

SUMMARY:
The preschool years are a critical time for shaping food preferences and eating behaviors, which affect dietary behaviors in adults and life-long risks for obesity, diabetes, cardiovascular disease, and other chronic conditions. Unfortunately, many US children, especially low-income and ethnic minorities, have dietary patterns associated with obesity and increased morbidity. Thus, to improve child diet quality, it is essential to develop effective targeted interventions in settings where children (especially higher-risk children) spend time. The investigators build upon our efficacious Healthy Start intervention with family childcare home (FCCH) providers (FCCP) to pilot a novel, 8-month multilevel tailored intervention to reach families through FCCH. This would be the first study to incorporate family-based intervention components into FCCH. The 8-month intervention will include an adapted version of the Healthy Start intervention as well as FCCP training to deliver nutrition messages to parents using an existing childcare App, complemented with FCCH environmental cues and tailored print and videos for parents. In sum, feasible and effective interventions to improve young children's diets are urgently needed. The FCCH is a novel and untapped setting to intervene with both FCCP and parents simultaneously to affect children's diets in both childcare and home settings, which has the potential to more fully impact the child's overall diet and weight status.

DETAILED DESCRIPTION:
The preschool years are a critical time for shaping food preferences and eating behaviors which, in turn, affect dietary behaviors in adults and life-long risks for obesity, diabetes, cardiovascular disease and other chronic conditions. Unfortunately, many US children, especially low-income and ethnic minorities, have dietary patterns associated with obesity and increased morbidity. Thus, to improve child diet quality, it is essential to develop effective targeted interventions in settings where children (especially higher risk children) spend time. There is a national call for dietary interventions that span multiple settings including the childcare and home environments. In response to PAS-20-160, the investigators build upon our efficacious Healthy Start intervention with family childcare home (FCCH) providers (FCCP) to pilot a novel, 8-month multilevel tailored intervention to reach families through FCCH. This would be the first study to incorporate family-based intervention components into FCCH. FCCH are a promising intervention setting as parents trust FCCPs as extended family members and FCCP feel comfortable talking to parents about children's diet, but want more training to do so effectively. The 8-month intervention will include an adapted version of the Healthy Start intervention for English and Spanish-speaking FCCP as well as FCCP training to deliver nutrition messages to parents using an existing childcare App, complemented with FCCH environmental cues and tailored print and videos for parents. Specific Aims are to: SA.1. Conduct formative research with FCCP and parents to inform refinement of the multi-level intervention. SA.2. Conduct a pilot trial with 40 FCCP and 80 parents with 18-54-month-old children to evaluate feasibility and acceptability of intervention and study protocols, and preliminary efficacy of the nutrition intervention compared to an attention-matched control on: a). children's dietary quality at FCCH and home, b). social/physical FCCH and home food environments, c). children's dermal carotenoid levels and z-BMI scores. SA3. Conduct post qualitative interviews with parents, FCCP, coaches, staff & partners to assess the intervention's acceptability and suggestions for improvement. In sum, feasible and effective interventions to improve young children's diets are urgently needed. The FCCH is a novel and untapped setting to intervene with both FCCP and parents simultaneously to affect children's diets in both the childcare and home settings, which has the potential to more fully impact the child's overall diet and weight status. This pilot feasibility research of a novel, multi-level intervention will inform a future full-scale cluster RCT, which will fill important research gaps and move the frontier of nutrition research forward.

ELIGIBILITY:
Providers:

Inclusion Criteria:

* English and/or Spanish-speaking and reading
* State licensed family childcare providers (FCCP)
* FCCP that care for 18-54 month-old children,
* Plan for FCCH to be in operation for the next year
* Willing to be randomized to either study arm,
* Have at least 2 eligible children in their care with at least 1 parent-child dyad consenting to participate

Exclusion Criteria:

* Participation in the prior Healthy Start Project

Parents:

Inclusion Criteria:

* English and/or Spanish-speaking and reading
* Legal guardian of child(ren) who receive care in a participating FCCH
* Child(ren) must be 18-54 months-old
* Care must be for at least 15 hrs./wk
* Plan to continue childcare with their current FCCP for the next 9 months
* Be the caregiver mainly responsible for the child's eating at home
* Willing to be randomized (with the FCCP) to either study arm

Exclusion Criteria:

* Not meeting above criteria.

Children:

Inclusion Criteria:

* Children 18-54 months-old who receive care in a participating FCCH
* Care must be for at least 15 hours per week
* Agree to be measured (All other evaluation is observation that does not require assent).

Exclusion Criteria:

- Not meeting above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Score | 9 Months
  Feasibility Score Recruitment and retention success will be measured and scored. Higher scores will indicate higher recruitment and retention.
Acceptability Score | 9 months
  Acceptability Score Participant providers and parents rate the intervention as acceptable, which will be coded as a score. Higher score will indicate higher acceptability of the intervention.
Child diet at home | Baseline and 9 months
  HEI Score - Diet Quality at Home Parents will be called on two randomly selected days (at least one weekend day) and asked to recall child's food intake in previous 24-hours using gold standard multiple-pass method. Parents will report child's foods and beverage intake on the previous day (excluding child intake while outside their care) using established methods as in our Healthy Start diversity supplement. Data will be entered into the NDSR program, which will be used to average data across both days and then calculate HEI-2015 score using same methods as for childcare.
Dietary Observation in Child Care | Baseline and 9 months
  HEI Score - Diet Quality in Childcare Dietary Observation for Childcare (DOCC) is a validated visual observation technique that minimizes observer intrusion, so children don't know intake is being observed. Observers visually estimate and record amount /type of foods/beverages served to children in meals/snacks. Foods not easily discerned will be clarified with FCCP (e.g. food prep, brand names). Amount of food wasted (e.g. dropped, spilled, traded) and remaining will be recorded and amount of food consumed will be estimated as amount served - amount remaining. -Both days of observation data will be entered into NDSR, and averaged to estimate daily nutrient and food data. -Nutrient content, HEI-2015 total and component scores will be derived

SECONDARY OUTCOMES:
Veggie Meter | Baseline and 9 months
  Carotenoid Score Provides an objective measure of F&V intake using reflection spectroscopy to detect non-invasively, the level of carotenoids in the child's skin.
Environment and Policy Assessment and Observation Tool | Baseline and 9 months
  EPAO Score Measures childcare nutrition environments and practices over a full-day.
Child Weight | Baseline and 9 months
  Weight (kg) Investigators will use standard techniques for measuring child weight in kilograms
Child Height | Baseline and 9 months
  Height (cm) Investigators will use standard techniques for measuring child height in cm.
Feeding Practices | Baseline and 9 months
  CFPQ Score Parents will be surveyed about their feeding practices of their own children at home. 32 questions from the Comprehensive Feeding Practices Questionnaire (CFPQ) will be used.
Beverage Intake Questionnaire (BEVQ-PS) | Baseline and 9 months
  BEVQ-PS is a valid instrument used to assess SSB, water, and whole-milk intake.
Rapid Prime Diet Quality Score (rPDQS) | Baseline and 9 months
  rPDQS Score The rPDQS is a valid, brief diet quality screener that identifies clinically relevant patterns of food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M Risica, DrPH, Principal Investigator — Brown School of Public Health

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This information will be available for five years after the completion of the main effects papers.
Access Criteria: Contact one of the MPIs for access.

REFERENCES:
- [Background] Gans KM, Tovar A, Kang A, Ward DS, Stowers KC, von Ash T, Dionne L, Papandonatos GD, Mena N, Jiang Q, Risica PM. A multi-component tailored intervention in family childcare homes improves diet quality and sedentary behavior of preschool children compared to an attention control: results from the Healthy Start-Comienzos Sanos cluster randomized trial. Int J Behav Nutr Phys Act. 2022 Apr 15;19(1):45. doi: 10.1186/s12966-022-01272-6. PMID 35428298
- [Background] Risica PM, Tovar A, Palomo V, Dionne L, Mena N, Magid K, Ward DS, Gans KM. Improving nutrition and physical activity environments of family child care homes: the rationale, design and study protocol of the 'Healthy Start/Comienzos Sanos' cluster randomized trial. BMC Public Health. 2019 Apr 18;19(1):419. doi: 10.1186/s12889-019-6704-6. PMID 30999881
- [Background] Tovar A, Risica PM, Ramirez A, Mena N, Lofgren IE, Cooksey Stowers K, Gans KM. Exploring the Provider-Level Socio-Demographic Determinants of Diet Quality of Preschool-Aged Children Attending Family Childcare Homes. Nutrients. 2020 May 11;12(5):1368. doi: 10.3390/nu12051368. PMID 32403299
- [Background] Ramirez A, Vadiveloo M, Risica PM, Gans KM, Greaney ML, Mena NZ, Cooksey Stowers K, Tovar A. Dietary Contributors to Food Group Intake in Preschool Children Attending Family Childcare Homes: Differences between Latino and Non-Latino Providers. Nutrients. 2020 Nov 29;12(12):3686. doi: 10.3390/nu12123686. PMID 33260442
- [Background] Jiang Q, Risica PM, Tovar A, Stowers KC, Schwartz MB, Lombardi C, Gans KM. Mediation of the Association between Social Environmental Characteristics of Family Childcare Home and Weight Status in Children by Diet Quality. Res Sq [Preprint]. 2023 Aug 16:rs.3.rs-3147729. doi: 10.21203/rs.3.rs-3147729/v1. PMID 37645722
- [Background] Jiang Q, Risica PM, Tovar A, Stowers KC, Schwartz MB, Lombardi C, Alhassan S, Gans KM. Effect of Applying Best Practices for Physical Activity and Screen Time to Family Childcare Homes. Prev Chronic Dis. 2023 Jul 13;20:E60. doi: 10.5888/pcd20.220325. PMID 37441753
- [Background] Jiang Q, Tovar A, Risica PM, Cooksey Stowers K, Schwartz M, Lombardi C, Kang A, Mena NZ, Gans KM. Ethnic Differences in Family Childcare Providers' Nutrition- and Activity-Related Attitudes and Barriers. J Obes. 2021 Oct 7;2021:6697006. doi: 10.1155/2021/6697006. eCollection 2021. PMID 34659829